CLINICAL TRIAL: NCT04051775
Title: Non-Pharmacological Treatment of Psychosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/938
Record Dates: First submitted 2019-05-16; First posted 2019-08-09 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-07

CONDITIONS: Psychosis; Schizophrenia-Like
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectives of the project are to investigate feasibility, safety, and health-related outcomes in patients with psychosis who choose not to use antipsychotic drugs (APs). The instruction from the Ministry of Health and Care Services to establish "Medication Free" (non-pharmacological (NonPharm)) treatment services, which has received substantial critique for being given without support in scientific evidence, provides a window of opportunity for research in an under-investigated field. The study will prospectively follow a cohort over 1 year who seeks NonPharm treatment, with repeated measurements of symptoms, functional outcomes, quality of life, adverse events, as well as biological parameters including genetics and brain imaging, and environmental factors, and compare the findings to a control group of users of antipsychotic drugs, matched for age, gender and diagnosis. Current unanswered questions in the treatment of psychosis include which patients can successfully and safely discontinue antipsychotic medication; and what are the long-term symptomatic, biological and functional outcomes after use or non-use of APs, respectively. Taken together there is a fundamental lack of high-quality evidence to guide the treatment options in people who cannot or do not want to use APs in psychosis. This is also a major challenge in the study, as a more rigorous design that could directly compare different treatment options is not feasible, because no alternatives to APs have proven to be sufficiently effective and safe in controlled trials. The study is accordingly expected to provide new exploratory information that could be the basis of intervention studies which in its turn could provide important information for consumers and the mental health services regarding treatment options in psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of diagnostic criteria for schizophrenia or related disorder (corresponding to chapter F2 in the ICD-10)
* The clinician responsible for the treatment must consider nonpharmacological treatment to be professionally justifiable in the patient in question
* Patient being able/ capable of providing informed consent
* Patient receiving active treatment including different psychosocial treatments
* Patient having a treatment plan and a crisis resolution plan.

Exclusion Criteria Not fullfilling inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients are those seeking NonPharm treatment who has a diagnosis of schizophrenia or related disorder (corresponding to chapter F2 in the ICD-10). Eligible patients will be included from the Division of Psychiatry, Haukeland University Hospital and collaborating District Psychiatric Centers in the same catchment area. The catchment population is 400.000. Both in- and out-patients are eligible for the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Serious adverse events | One year
  To investigate the prevalence of any Serious Adverse Events (SAE) in the NorPharm group compared to the control group

SECONDARY OUTCOMES:
Time to remission | One year
  To investigate the time to remission (absence of positive psychotic symptoms as determined by the Positive And Negative Syndrome Scale)
Time to recovery | One year
  To investigate the time to recovery (absence of positive psychotic symptoms plus normalized functioning)
Time to relapse | One year
  To investigate the time to relapse (presence of positive psychotic symptoms)
Insight | One year
  To investigate the change of insight as determined by Beck Cognitive Insight Scale (BCIS)
Insight | One year
  To investigate the change of insight as determined by Medication Adherence Report Scale
Insight | One year
  To investigate the change of insight as determined by Birchwood Insight Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland Univsersity Hospital, Bergen, Norway